CLINICAL TRIAL: NCT03719170
Title: Evaluation of the National Randomized Proton Pump Inhibitor De-prescribing (RaPPID) Program
Acronym: RaPPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 18-151
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-04

CONDITIONS: Proton Pump Inhibitors
Keywords: proton pump inhibitors; program evaluation; low-value care; de-implementation; patient safety

STUDY DESIGN:
Intervention Model Description: A cluster-randomized (by Veterans Integrated Service Networks or VISN) pragmatic trial of the provider-centered intervention versus pragmatic control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- De-prescribing Program (Experimental): The 9 Veterans Integrated Service Networks (VISNs) randomly assigned to the PPI de-prescribing program. VISNs are the 18 geographical regions that make up the VHA.
  PPI De-prescribing Program: The PPI de-prescribing program included alerts to clinical pharmacy specialists and primary care providers informing them of individual patients scheduled for upcoming primary care visits who meet criteria for PPI de-prescription; activation of clinical pharmacy specialists; education of primary care providers; and patient education.
  Interventions: Behavioral: PPI De-prescribing Program
- No De-prescribing Program (No Intervention): The 8 Veterans Integrated Service Networks (VISNs) randomly assigned to usual care and did not receive the national de-prescribing program. VISNs are the 19 geographical regions that make up the VHA.

INTERVENTIONS:
Behavioral: PPI De-prescribing Program — The PPI de-prescribing program includes alerts to clinical pharmacy specialists and primary care providers informing them of individual patients scheduled for upcoming primary care visits who meet criteria for PPI de-prescription; activation of clinical pharmacy specialists; education of primary care providers; and patient education.
  Other Names: RaPPID
  Arms: De-prescribing Program

SUMMARY:
Proton pump inhibitors (PPIs) are medications used to treat acid-related stomach disorders, such as chronic heartburn. These medications are widely used by Veterans, with over 11 million 30-day prescriptions being filled each year. Though they are highly effective, long-term use of PPIs may be harmful. For this reason, experts recommend that PPIs be stopped in patients who do not have a clear need for these medications. Unfortunately, PPIs continue to be overused. To address this issue, the VA is implementing a national program to de-prescribe (i.e., reduce the dose of, or stop) PPIs. In this study, the investigators will be evaluating this national program by assessing: (a) how successfully the program was implemented; (b) understanding how effective the program was in improving appropriate use of PPIs; and, (c) ensuring no unintended consequences (such as peptic ulcer bleeding) occurred with PPI de-prescribing. This study addresses a potential safety concern for Veterans and aligns with VA's broader goal of de-implementing low-value care.

DETAILED DESCRIPTION:
Background: Proton pump inhibitors (PPIs) are among the most commonly prescribed medications in the Veterans Health Administration (VHA), accounting for over 11 million 30-day prescriptions and nearly $50 million in medication costs annually. Though effective for treatment of acid-related disorders such as gastroesophageal reflux disease, PPIs have been associated with a number of potential harms in observational studies (e.g., dementia, chronic kidney disease, fractures), and increased mortality in Veterans. Nonetheless, PPIs continue to be used without an appropriate indication or for longer and at higher doses than necessary. Accordingly, VHA Pharmacy Benefits Management Services (PBM) will deploy RaPPID - a national Randomized PPI De-prescribing program - in Fiscal Year 2018 targeting patients for whom a short course of PPI is likely sufficient. This program will comprise activation of Clinical Pharmacy Specialists, provider education and academic detailing, and patient education. In partnership with PBM, the investigators propose to conduct an evaluation of this national program in a cluster-randomized design.

Objectives: (1) assess the impact of the de-prescribing program on important clinical outcomes, and to understand how and why these outcomes were achieved or not achieved (outcomes and process evaluation); (2) assess the economic effects of the de-prescribing program (economic evaluation).

Methods: The investigators will then assess the impact of RaPPID on PPI use (primary outcome) in a cluster randomized design (cluster = Veterans Integrated Service Network (VISN). The investigators will also assess a variety of unintended effects, including impact of reduced PPI use on upper GI symptoms and complications such as upper GI bleeding. Furthermore, the investigators will use process evaluation approaches to understand why and how the program was effective or ineffective in specific contexts. Finally, the investigators will use data from the outcomes evaluation of this proposal to estimate the budget impact of RaPPID, taking into account the impact of the program on VHA and non-VHA healthcare utilization.

Impact: RaPPID will be among the largest concerted efforts at de-prescribing ever undertaken in VHA. Prospective evaluation of the program therefore presents a unique opportunity not only to enhance the program itself, but also to gain insights about how to reduce the use of low-value services more broadly, a key VHA priority for the coming decade. Importantly, the prospective, controlled study design the investigators propose will also allow us to make strong claims about whether PPIs cause the putative adverse effects to which they have been linked. Ultimately, this evaluation will provide not only valuable insight into the benefits and harms of a national effort to appropriately de-prescribe PPIs, but also broader lessons about how to effectively undertake other such interventions to de-implement entrenched clinical practices in the future.

ELIGIBILITY:
Inclusion Criteria:

Chronic PPI users defined as 90-day prescription during the 120-day period prior to a scheduled VA primary care visit who receive:

1. Once-daily PPI with

   * No clear indication for PPIs, OR
   * Uncomplicated Gastroesophageal reflux disease (GERD) OR
2. Twice-daily PPI for any indication except Zollinger-Ellison

Exclusion Criteria:

Patients taking once-daily PPIs will be excluded if they have one or more of the following characteristics:

* Eosinophilic esophagitis
* Esophagitis
* Esophageal ulcer
* Esophageal stenosis/stricture
* Dysphagia (other than oropharyngeal)
* Barrett's esophagus
* Peptic ulcer
* Zollinger-Ellison
* Idiopathic pulmonary fibrosis
* NSAID + age > 65 yrs, 2nd NSAID, aspirin, anti-thrombotic, OR corticosteroid
* Aspirin + age 60 yrs, NSAID, anti-thrombotic, OR corticosteroid
* Pancreatic enzyme replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220306 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer D. Saini, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (4):
- United States (4):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spechler SJ, Hunter JG, Jones KM, Lee R, Smith BR, Mashimo H, Sanchez VM, Dunbar KB, Pham TH, Murthy UK, Kim T, Jackson CS, Wallen JM, von Rosenvinge EC, Pearl JP, Laine L, Kim AW, Kaz AM, Tatum RP, Gellad ZF, Lagoo-Deenadayalan S, Rubenstein JH, Ghaferi AA, Lo WK, Fernando RS, Chan BS, Paski SC, Provenzale D, Castell DO, Lieberman D, Souza RF, Chey WD, Warren SR, Davis-Karim A, Melton SD, Genta RM, Serpi T, Biswas K, Huang GD. Randomized Trial of Medical versus Surgical Treatment for Refractory Heartburn. N Engl J Med. 2019 Oct 17;381(16):1513-1523. doi: 10.1056/NEJMoa1811424. PMID 31618539
- [Result] Kurlander JE, Rubenstein JH, Richardson CR, Krein SL, De Vries R, Zikmund-Fisher BJ, Yang YX, Laine L, Weissman A, Saini SD. Physicians' Perceptions of Proton Pump Inhibitor Risks and Recommendations to Discontinue: A National Survey. Am J Gastroenterol. 2020 May;115(5):689-696. doi: 10.14309/ajg.0000000000000558. PMID 32091419
- [Result] Simonov M, Abel EA, Skanderson M, Masoud A, Hauser RG, Brandt CA, Wilson FP, Laine L. Use of Proton Pump Inhibitors Increases Risk of Incident Kidney Stones. Clin Gastroenterol Hepatol. 2021 Jan;19(1):72-79.e21. doi: 10.1016/j.cgh.2020.02.053. Epub 2020 Mar 6. PMID 32147588
- [Result] Laine L. Colonoscopy for Lower Gastrointestinal Bleeding-Time Is Not of the Essence. Gastroenterology. 2020 Jan;158(1):38-39. doi: 10.1053/j.gastro.2019.11.009. Epub 2019 Nov 12. No abstract available. PMID 31730767
- [Result] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Result] Saffouri E, Blackwell C, Laursen SB, Laine L, Dalton HR, Ngu J, Shultz M, Norton R, Stanley AJ. The Shock Index is not accurate at predicting outcomes in patients with upper gastrointestinal bleeding. Aliment Pharmacol Ther. 2020 Jan;51(2):253-260. doi: 10.1111/apt.15541. Epub 2019 Oct 23. PMID 31642558
- [Result] Laine L. Timing of Endoscopy in Patients Hospitalized with Upper Gastrointestinal Bleeding. N Engl J Med. 2020 Apr 2;382(14):1361-1363. doi: 10.1056/NEJMe2002121. No abstract available. PMID 32242363
- [Result] Lee MW, Pourmorady JS, Laine L. Use of Fecal Occult Blood Testing as a Diagnostic Tool for Clinical Indications: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2020 May;115(5):662-670. doi: 10.14309/ajg.0000000000000495. PMID 31972617
- [Result] Campbell EV 3rd, Muniraj T, Aslanian HR, Laine L, Jamidar P. Musculoskeletal Pain Symptoms and Injuries Among Endoscopists Who Perform ERCP. Dig Dis Sci. 2021 Jan;66(1):56-62. doi: 10.1007/s10620-020-06163-z. Epub 2020 Mar 6. PMID 32144599
- [Result] Shung D, Laine L. Machine Learning Prognostic Models for Gastrointestinal Bleeding Using Electronic Health Record Data. Am J Gastroenterol. 2020 Aug;115(8):1199-1200. doi: 10.14309/ajg.0000000000000720. PMID 32530828
- [Result] Laursen SB, Oakland K, Laine L, Bieber V, Marmo R, Redondo-Cerezo E, Dalton HR, Ngu J, Schultz M, Soncini M, Gralnek I, Jairath V, Murray IA, Stanley AJ. ABC score: a new risk score that accurately predicts mortality in acute upper and lower gastrointestinal bleeding: an international multicentre study. Gut. 2021 Apr;70(4):707-716. doi: 10.1136/gutjnl-2019-320002. Epub 2020 Jul 28. PMID 32723845
- [Result] Kelly CR, Laine LA, Wu GD. Monitoring Fecal Microbiota Transplantation Practice in a Rapidly Evolving Health and Regulatory Environment. Gastroenterology. 2020 Dec;159(6):2004-2006. doi: 10.1053/j.gastro.2020.08.039. Epub 2020 Aug 22. No abstract available. PMID 32841646
- [Result] Vyas M, Celli R, Singh M, Patel N, Aslanian HR, Boffa D, Deng Y, Ciarleglio MM, Laine L, Jain D. Intestinal metaplasia around the gastroesophageal junction is frequently associated with antral reactive gastropathy: implications for carcinoma at the gastroesophageal junction. Hum Pathol. 2020 Nov;105:67-73. doi: 10.1016/j.humpath.2020.08.007. Epub 2020 Sep 14. PMID 32941964
- [Result] Kurlander JE, Barnes GD, Sukul D, Helminski D, Kokaly AN, Platt K, Gurm H, Saini SD. Trials of Dual Antiplatelet Therapy After Percutaneous Coronary Intervention Lack Strategies to Ensure Appropriate Gastroprotection. Am J Gastroenterol. 2021 Apr;116(4):821-824. doi: 10.14309/ajg.0000000000001134. PMID 33982954
- [Result] Targownik LE, Fisher DA, Saini SD. AGA Clinical Practice Update on De-Prescribing of Proton Pump Inhibitors: Expert Review. Gastroenterology. 2022 Apr;162(4):1334-1342. doi: 10.1053/j.gastro.2021.12.247. Epub 2022 Feb 17. PMID 35183361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a national Veterans Health Administration (VHA) program. Randomization was at the level of geographical regions called Veterans Integrated Service Networks (VISNs). At the date of randomization (8/27/2019), there were 18 VISNs. One VISN was excluded because it was the model for the national program. Out of 17 VISNs, 8 were randomized to the control arm and 9 to the intervention arm. Subjects were identified via an electronic algorithm during the recruitment year 9/16/2019 - 9/15/2020.
Units Other Than Participants: VA regional delivery network (VISN)
Groups:
- De-prescribing Program: The 9 Veterans Integrated Service Networks (VISNs) randomly assigned to the Proton Pump Inhibitor (PPI) de-prescribing program. VISNs are the 18 geographical regions that make up the VHA.
  PPI De-prescribing Program: The PPI de-prescribing program included alerts to clinical pharmacy specialists and primary care providers informing them of individual patients scheduled for upcoming primary care visits who meet criteria for PPI de-prescription; activation of clinical pharmacy specialists; education of primary care providers; and patient education.
- No De-prescribing Program: The 8 Veterans Integrated Service Networks (VISNs) randomly assigned to usual care and did not receive the national de-prescribing program. VISNs are the 18 geographical regions that make up the VHA.
Period: Overall Study
Arm/Group | De-prescribing Program | No De-prescribing Program
Started | 119494; 9 VA regional delivery network (VISN) | 100812; 8 VA regional delivery network (VISN)
Completed | 119494; 9 VA regional delivery network (VISN) | 100812; 8 VA regional delivery network (VISN)
Not Completed | 0; 0 VA regional delivery network (VISN) | 0; 0 VA regional delivery network (VISN)

BASELINE CHARACTERISTICS:
Groups:
- No De-prescribing Program: The 8 Veterans Integrated Service Networks (VISNs) randomly assigned to usual care and will not receive the national de-prescribing program. VISNs are the 18 geographical regions that make up the VHA.
- Total: Total of all reporting groups
Arm/Group | De-prescribing Program | No De-prescribing Program | Total
Number analyzed (Participants) | 119,494 | 100,812 | 220306
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.74 (13.00) | 64.63 (13.19) | 64.69 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants] — Data were collected via algorithm from electronic health records. Population: Row population differs from the Overall because 10 participants had missing Sex data: 4 from the De-prescribing Program arm and 6 from the No De-prescribing Program arm.
  Participants
    Sex: number analyzed (Participants) | 119,490 | 100,806 | 220296
    Sex: Female | 8,101 | 7,036 | 15137
    Sex: Male | 111,389 | 93,770 | 205159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2,624 | 7,757 | 10381
  Not Hispanic or Latino | 116,866 | 93,049 | 209915
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 825 | 785 | 1610
  Asian | 716 | 547 | 1263
  Native Hawaiian or Other Pacific Islander | 816 | 669 | 1485
  Black or African American | 16,964 | 13,948 | 30912
  White | 93,976 | 79,990 | 173966
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6,197 | 4,873 | 11070
Charlson Comorbidity Index (CCI) [Count of Participants; unit: Participants] — Measure of overall health state, with lower score indicating better health and higher score indicating worse health, assessed electronically. For further details, see Charlson, ME. Psychother Psychosom. 2022;91(1):8-35.
  Participants
    Charlson Comorbidity Index = 0 | 44,970 | 37,710 | 82680
    Charlson Comorbidity Index = 1 | 30,391 | 24,781 | 55172
    Charlson Comorbidity Score = 2 | 14,889 | 12,598 | 27487
    Charlson Comorbidity Index = 3 | 11,982 | 10,312 | 22294
    Charlson Comorbidity Index = 4 | 6,329 | 5,412 | 11741
    Charlson Comorbidity Index >= 5 | 10,933 | 9,999 | 20932

OUTCOME MEASURES:

1. Primary Outcome: PPI Prescribing (H1)
Description: The proportion of days proton pump inhibitors are prescribed in the 12 months following the index visit.
Time Frame: 12 months
Population: All participants from the 17 randomized VISNs meeting study criteria within the 1-year recruitment period.
Measure: Mean (Standard Deviation); unit: percentage of days on PPI
Groups:
- No De-prescribing Program: The 8 Veterans Integrated Service Networks (VISNs) randomly assigned to usual care and which did not receive the national de-prescribing program. VISNs are the 18 geographical regions that make up the VHA.
Arm/Group | De-prescribing Program | No De-prescribing Program
Number analyzed (Participants) | 119494 | 100812
percentage of days on PPI | 73.69 (0.27) | 72.66 (0.27)
Statistical Analysis 1: Comparison: De-prescribing Program vs No De-prescribing Program; Power Calculation: Assuming approximately the same number of eligible subjects in each VISN (with an average of 10,563 candidates per VISN) and an Intraclass correlation coefficient (ICC) of 0.12, randomizing 17 VISNs will give more than 80% power to detect % days on PPI of 75% vs. 50%, 85% vs. 60%, 80% vs. 55%, or 70% vs. 45%, but to detect a difference between 70% vs. 50%, power is only 61% using 0.05 level 2-sided test; Test type: Superiority; Slope = 0.0000684, 95% CI 2-sided [-0.0003 to 0.000413]

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assessed. Specifically, because this was a minimal risk study with no intervention (i.e., program evaluation), involving use of electronic data, paper and telephone surveys, and telephone interviews about PPI de-prescribing experiences.
Groups:
- De-prescribing Program: Veterans Integrated Service Networks (VISNs) randomly assigned to the PPI de-prescribing program. VISNs are the 19 geographical regions that make up the VHA.
  PPI De-prescribing Program: The PPI de-prescribing program includes alerts to clinical pharmacy specialists and primary care providers informing them of individual patients scheduled for upcoming primary care visits who meet criteria for PPI de-prescription; activation of clinical pharmacy specialists; education of primary care providers; and patient education.
- No De-prescribing Program: Veterans Integrated Service Networks (VISNs) randomly assigned to usual care and will not receive the national de-prescribing program. VISNs are the 19 geographical regions that make up the VHA.
Arm/Group | De-prescribing Program | No De-prescribing Program
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The following issues likely contributed to decreased implementation of intervention:

1. Ranitidine was a key "step down" medication to use in place of PPIs, but a national shortage disrupted its availability; and,
2. COVID-19 pandemic 6 months into intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03719170/Prot_SAP_000.pdf